CLINICAL TRIAL: NCT05404659
Title: Comparative Effects of Oscillatory Mobilizations and Mckenzie Retraction Exercises on Pain, Range of Motion and Disability in Patients With Mechanical Neck Pain
Brief Title: Comparative Effects of Oscillatory Mobilizations and Mckenzie Retraction Exercises on Mechanical Neck Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR&AHS/22/0124
Record Dates: First submitted 2022-05-31; First posted 2022-06-03 (Actual); Last update posted 2022-06-03 (Actual); Status verified 2022-05

CONDITIONS: Mechanical Neck Pain
Keywords: Cervical spine; exercise therapy; pain; Manual therapy
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Oscillatory Mobilizations (Active Comparator)
  Interventions: Other: Oscillatory Mobilization
- Mckenzie Retraction Exercises (Experimental)
  Interventions: Other: Mckenzie Retraction Exercises

INTERVENTIONS:
Other: Oscillatory Mobilization — conventional physical therapy treatment, postural correction and maitland's oscillatory mobilizitions.
  Arms: Oscillatory Mobilizations
Other: Mckenzie Retraction Exercises — conventional physical therapy treatment, postural correction and Mckenzie retraction exercises.
  Arms: Mckenzie Retraction Exercises

SUMMARY:
The neck pain is a public health problem and a common source of disability in the general population. Its exact pathology remains obscure, but the source of symptoms has been asserted to involve mechanical dysfunction of the cervical spine, particularly the zygoapophysial joints. Among the diversity of neck pain, mechanical neck pain is the most common type, with the pain primarily confined in the area on the posterior aspect of the neck that can be exacerbated by neck movements or by sustained neck postures. The usual clinical presentation of this mechanical neck pain is a reduction in mobility of either a single segment or multiple segments of the cervical spine in association with pain. This study will be a randomized control trial and will be conducted at Arif Memorial Teaching Hospital Lahore. The study will be completed within the time duration of six months. Convenience sampling technique will be used to collect data. A sample size of 30 patients(15 in each group) which will fulfill inclusion criteria will be taken in the study. Participants will be divided into two groups. Both Groups will be given conventional physical therapy and postural correction education. Group A will be provide oscillatory mobilizations. The following grades will be use: grades I and II for pain and grades III and IV to increase joint range of motion. This oscillatory mobilization will perform at a rate of 2-3 oscillations per second. and a frequency of 3-4 mobilization of the joint lasting approximately 30 sec each.

The rest time between each mobilization will be one minute for 5 days a week for four weeks , while group B will be treat withmckenzie retraction exercises in which foursets of 10-15 repetitions with 1-2 minutes rest between each set for 5 days a week during four weeks. Data will collect by using tools like numeric pain rating scale to measure pain, universal goniometer will be use for range of motion and disability level will be record pre and post treatment by using neck disability index. Then data will analyzed by using SPSS.

ELIGIBILITY:
Inclusion Criteria:

Patient with primary complaint of non specific neck pain. Pain of sufficient intensity (greater than 2 out of 10 on numerical pain scale) · Pain and stiffness for at least 2 weeks Pain aggravated by neck movement ·

Exclusion Criteria:

History of orthopedic surgery to the neck and shoulder and Temporo-mandibular Joint neurological symptoms due to cervical dysfunction History of Carcinoma Progressive neurological deficits

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 26 (Estimated)
Dates: Start 2022-05-25 (Estimated); Primary Completion 2022-10-25 (Estimated); Study Completion 2023-01-25 (Estimated)

PRIMARY OUTCOMES:
Neck pain | 5 week
  Numeric pain rating scale is valid and reliable tool to measure pain
Range of motion | 5 week
  Goniometre is used to measure ROM. It measurement has been found to have greater intra-tester reliability in both clinical and research settings
Disability | 5 week
  The Neck Disability Index is the most widely used instrument for assessing self-rated disability in patients with neck pain

CONTACTS AND LOCATIONS:
Overall Officials: Saba Rafique, Phd*, Principal Investigator — Riphah International University
Locations (1):
- Arif Memorial Teaching Hospital, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Osama M, Shakil Ur Rehman S. Effects of static stretching as compared to autogenic inhibition and reciprocal inhibition muscle energy techniques in the management of mechanical neck pain: a randomized controlled trial. J Pak Med Assoc. 2020 May;70(5):786-790. doi: 10.5455/JPMA.9596. PMID 32400728
- [Background] Hassan F, Osama M, Ghafoor A, Yaqoob MF. Effects of oscillatory mobilization as compared to sustained stretch mobilization in the management of cervical radiculopathy: A randomized controlled trial. J Back Musculoskelet Rehabil. 2020;33(1):153-158. doi: 10.3233/BMR-170914. PMID 31127753
- [Background] Shabbir M, Arshad N, Naz A, Saleem N. Clinical outcomes of maitland mobilization in patients with Myofascial Chronic Neck Pain: A randomized controlled trial. Pak J Med Sci. 2021 Jul-Aug;37(4):1172-1178. doi: 10.12669/pjms.37.4.4220. PMID 34290803
- [Background] Raja G P, Bhat N S, Fernandez-de-Las-Penas C, Gangavelli R, Davis F, Shankar R, Prabhu A. Effectiveness of deep cervical fascial manipulation and yoga postures on pain, function, and oculomotor control in patients with mechanical neck pain: study protocol of a pragmatic, parallel-group, randomized, controlled trial. Trials. 2021 Aug 28;22(1):574. doi: 10.1186/s13063-021-05533-w. PMID 34454582
- [Background] Young IA PT, DSc, Dunning J PT, DPT, Butts R PT, PhD, Mourad F PT, DPT, Cleland JA PT, PhD. Reliability, construct validity, and responsiveness of the neck disability index and numeric pain rating scale in patients with mechanical neck pain without upper extremity symptoms. Physiother Theory Pract. 2019 Dec;35(12):1328-1335. doi: 10.1080/09593985.2018.1471763. Epub 2018 Jun 1. PMID 29856244
- [Background] Kanlayanaphotporn R, Chiradejnant A, Vachalathiti R. The immediate effects of mobilization technique on pain and range of motion in patients presenting with unilateral neck pain: a randomized controlled trial. Arch Phys Med Rehabil. 2009 Feb;90(2):187-92. doi: 10.1016/j.apmr.2008.07.017. PMID 19236972
- [Background] Osama M, Tassadaq N, Malik RJ. Effect of muscle energy techniques and facet joint mobilization on spinal curvature in patients with mechanical neck pain: A pilot study. J Pak Med Assoc. 2020 Feb;70(2):344-347. doi: 10.5455/JPMA.14189. PMID 32063632
- [Background] Buyukturan O, Buyukturan B, Sas S, Kararti C, Ceylan I. The Effect of Mulligan Mobilization Technique in Older Adults with Neck Pain: A Randomized Controlled, Double-Blind Study. Pain Res Manag. 2018 May 15;2018:2856375. doi: 10.1155/2018/2856375. eCollection 2018. PMID 29861800